CLINICAL TRIAL: NCT03273244
Title: Towards a Better Understanding of What Palliative Sedated Patients Experience: Linking Numbers to Experiences
Brief Title: Measuring Comfort During Palliative Sedation
Acronym: COMPAS
Status: Completed | Type: Observational
Sponsor: Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Stefaan Six, Principal Investigator, Vrije Universiteit Brussel
Other Study IDs: FWOAL768
Record Dates: First submitted 2017-08-28; First posted 2017-09-06 (Actual); Last update posted 2019-10-18 (Actual); Status verified 2019-10

CONDITIONS: Palliative Sedation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Device monitoring: NeuroSense monitoring and ANI monitoring
  Interventions: Device: NeuroSense monitoring and ANI monitoring

INTERVENTIONS:
Device: NeuroSense monitoring and ANI monitoring — From the start of palliative sedation, monitoring of EEG with NeuroSense device (WAVcns: Wavelet Anesthetic Value of the Central Nervous System) and ANI-monitoring (Analgesia Nociception Index) will be initiated.

SUMMARY:
Background. In case of untreatable suffering at the end of life, palliative sedation may be chosen to assure comfort by reducing the patient's level of consciousness. An important question here is whether such sedated patients are certainly completely free of pain. Because these patients cannot communicate anymore, caregivers have to rely on observation to assess the patient's comfort. Recently however, more sophisticated techniques from the neurosciences (fMRI, EEG) have shown that sometimes consciousness and pain is undetectable with these traditional behavioral methods.

Therefore there is an urgent need for a more reliable way of assessment by combining existing observational scales, subjective assessments of caregivers and family and neuroimaging techniques.

Aim. The aim of this study is to better understand how unconscious palliative sedated patients experience the last days of their life and to find out if they are really free of pain.

Methods In this study the investigators will observe 40 patients starting with initiation of palliative sedation until death.

Assessment of comfort based on behavioural observations will be related with the results from a NeuroSense monitor, an EEG-based brain monitor used for evaluation of the adequacy of anesthesia and sedation in the operating room and an ECG-based Analgesia Nociception Index (ANI) monitor, which informs about the comfort or discomfort condition of the organism, based on the parasympathetic tone (including calculation of ANI). Additionally, the researchers will investigate whether changes of these measures can be linked to changes in the patients' experience as observed by caregivers and relatives, especially in the last moments of life. An innovative and challenging aspect of this study is its qualitative approach, implying all the different types of data will be used to link "objective" and "subjective" data to achieve a holistic understanding of the study topics.

The following data will be collected:

* assessment of pain/comfort by the patients themselves before loss of consciousness due to deep continuous sedation (if possible) by scoring a Visual Analogue Scale (VAS)
* brain function monitoring (NeuroSense monitor)
* monitoring of parasympathetic tone (ANI monitor)
* assessment by caregivers on 3 VAS scales (different scales or 3 different caregivers?)
* relatives' perception of the quality of the dying process on 3 VAS scales (idem)
* assessment by 2 trained investigators using observational scales
* observation: video and audio registration

ELIGIBILITY:
Inclusion Criteria:

Patients may be included if they are considered by their treating physician as:

1. in their last week of life
2. in conditions that might, when not treated, cause high levels of distress
3. sedated
4. unable to communicate

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients older than 18 years where palliative sedation is expected to be initiated, regardless of underlying diseases.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2017-05-12 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Level of awareness | From date of enrollment until the date of death, on average less than 1 week.
  Level of awareness as measured by a NeuroSense monitor and expressed as the WAVcns index (Wavelet-based Anesthetic Value for Central Nervous System). The WAVcns is based on cortical EEG.
Level of pain and discomfort | From date of enrollment until the date of death, on average less than 1 week.
  Level of pain and discomfort as measured by an ANI-monitor and expressed by the analgesia nociception index (ANI). The ANI is based on HRV (heart rate variability).

SECONDARY OUTCOMES:
Pain | From date of enrollment until the date of death (on average less than 1 week), during routine care, at least twice a day.
  Visual analog score assessment by nurse
Awareness | From date of enrollment until the date of death (on average less than 1 week), during routine care, at least twice a day.
  Visual analog score assessment by nurse
Communication | From date of enrollment until the date of death (on average less than 1 week), during routine care, at least twice a day.
  Visual analog score assessment by nurse
Pain | From date of enrollment until the date of death (on average less than 1 week), during visit, once a day.
  Visual analog score assessment by family member
Awareness | From date of enrollment until the date of death (on average less than 1 week), during visit, once a day.
  Visual analog score assessment by family member
Communication | From date of enrollment until the date of death (on average less than 1 week), during visit, once a day.
  Visual analog score assessment by family member

CONTACTS AND LOCATIONS:
Overall Officials: Reginald Deschepper, PhD, Study Chair — Vrije Universiteit Brussel
Locations (2):
- Belgium (2):
  - Algemeen Ziekenhuis Sint-Blasius, Dendermonde, Oost-Vlaanderen
  - University Hospital, Brussels

REFERENCES:
- [Derived] Six S, Laureys S, Poelaert J, Mairesse O, Theuns P, Bilsen J, Deschepper R. Neurophysiological Assessments During Continuous Sedation Until Death Put Validity of Observational Assessments Into Question: A Prospective Observational Study. Pain Ther. 2021 Jun;10(1):377-390. doi: 10.1007/s40122-020-00214-z. Epub 2020 Nov 5. PMID 33151515
- [Derived] Six S, Laureys S, Poelaert J, Bilsen J, Theuns P, Deschepper R. Comfort in palliative sedation (Compas): a transdisciplinary mixed method study protocol for linking objective assessments to subjective experiences. BMC Palliat Care. 2018 Apr 18;17(1):62. doi: 10.1186/s12904-018-0316-2. PMID 29669562